CLINICAL TRIAL: NCT00997802
Title: Evaluation of Accuracy of Computed Tomographic Colonography (CTC) in the Diagnosis of Colorectal Tumors by Gastroenterologists and Radiologists With Computer-aided Detection (CAD): A Multicenter Study
Brief Title: Japanese National Computed Tomographic (CT) Colonography Trial
Acronym: JANCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Japanese CT Colonography Society (Other)
Responsible Party: Principal Investigator, Hiroyuki Yoshida, 3D Imaging Laboratory, Massachusetts General Hospital, Japanese CT Colonography Society
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UMIN000002097
Record Dates: First submitted 2009-10-18; First posted 2009-10-19 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Colonic Polyps; Colonic Neoplasms
Keywords: Computed Tomographic Colonography; Colonic Polyps; Colonic Neoplasms; Computer Aided Diagnosis
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms | interventions — Colonography, Computed Tomographic

ARMS (1):
- CT colonography and optical colonoscopy (Other)
  Interventions: Device: CT colonography and optical colonoscopy

INTERVENTIONS:
Device: CT colonography and optical colonoscopy — All patients will undergo CT colonography and optical colonoscopy.

SUMMARY:
The purpose of this study is to evaluate the sensitivity of computed tomographic colonography (CTC) in detecting colorectal polyps and cancers in 1,500 subjects at increased risk of colorectal cancer (CRC), using optical colonoscopy as the reference standard.

DETAILED DESCRIPTION:
The investigators will evaluate the sensitivity of CTC in detecting colorectal polyps and cancers (at least 6 mm in diameter) in 1,500 subjects at increased risk of colorectal cancer (CRC), using optical colonoscopy as the reference standard. The primary endpoint will be sensitivity in the detection of colorectal polyps and cancers that are at least 6 mm in diameter. The secondary endpoints will include specificity and predictive values in the detection of colorectal polyps and cancers.

This clinical study will also evaluate the differences of the detection accuracies between human readings with and without computer-aided detection (CAD) that automatically detects colonic lesions in CTC images and presents the detected lesions to the readers. This clinical study will also compare performance between radiologists and gastroenterologists in detecting colorectal lesions in CTC images.

All the CTC images and their interpretations, optical colonoscopy reports and images, and pathology reports of resected colorectal lesion will be prospectively collected from 12 Japanese hospitals participating in the trial. All patients' information will be completely anonymized at each site before any analysis of the data takes place.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who are eligible for optical colonoscopy.
* Aged 20 years or older.
* Major functions of organs of the subjects are in a good condition.
* Signed informed consent forms are obtained from the patients.

Exclusion Criteria:

* Known colorectal polyps or cancers at any site at the time of enrollment.
* Patients with inflammatory bowel disease.
* Fulfillment of clinical criteria for diagnosis of FAP or HNPCC (Amsterdam criteria).
* Serious medical conditions that may increase the risk of optical colonoscopy or are so severe that screening would have no benefit.
* Previous colorectal surgery.
* Gastric or intestinal stenosis, abdominal adhesions, bowel obstruction or perforation, toxic megacolon.
* Evidence of an increased risk in carrying out bowel preparation or CTC exams.
* Possibility of pregnancy.
* Optical colonoscopy or barium enema carried out within the last 3 years.
* Patients with psychological conditions that contraindicate colonoscopy or that make them irrelevant to participate in the trial.
* Iodine hypersensitivity.
* Severe thyroid disease.
* Claustrophobia.
* Severe deafness.
* Subjects whose eligibility for this clinical trial is not appropriate by other reasons.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1257 (Actual)
Dates: Start 2009-10; Primary Completion 2015-12-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
sensitivity in the detection of colorectal polyps and cancers in CTC | 1.5 years

SECONDARY OUTCOMES:
specificity and predictive values in the detection of colorectal polyps and cancers in CTC. | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Koichi Nagata, MD, PhD, Study Director — Japanese CTC Society
Locations (12):
- Japanese CTC Society, 3D imaging Laboratory, Massachusetts General Hospital, Boston, Massachusetts, United States
- Japan (11):
  - Otarukyokai Hospital, Otaru, Hokkaido
  - Tonan Hospital, Sapporo, Hokkaido
  - Hokkaido Social Insurance Hospital, Sapporo, Hokkaido
  - Hokkaido Gastroenterology Hospital, Sapporo, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Showa University Northern Yokohama Hospital, Yokohama, Kanagawa
  - Kamigoto Hospital, Kamigotō, Nagasaki
  - Kawasaki Medical School, Kurashiki, Okayama-ken
  - Hamamatsu South Hospital, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital, Shimono, Tochigi
  - Tokyo Women's Medical University Medical Center East, Arakawa-ku, Tokyo

REFERENCES:
- [Result] Nagata K, Endo S, Honda T, Yasuda T, Hirayama M, Takahashi S, Kato T, Horita S, Furuya K, Kasai K, Matsumoto H, Kimura Y, Utano K, Sugimoto H, Kato H, Yamada R, Yamamichi J, Shimamoto T, Ryu Y, Matsui O, Kondo H, Doi A, Abe T, Yamano HO, Takeuchi K, Hanai H, Saida Y, Fukuda K, Nappi J, Yoshida H. Accuracy of CT Colonography for Detection of Polypoid and Nonpolypoid Neoplasia by Gastroenterologists and Radiologists: A Nationwide Multicenter Study in Japan. Am J Gastroenterol. 2017 Jan;112(1):163-171. doi: 10.1038/ajg.2016.478. Epub 2016 Oct 25. PMID 27779195
- See also: Original Contributions — http://www.nature.com/ajg/journal/v112/n1/full/ajg2016478a.html